CLINICAL TRIAL: NCT06832735
Title: Health-related Quality of Life of Women with Polycystic Ovary Syndrome At Sohag University Hospital
Status: Not yet recruiting | Type: Observational
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Samah Wagdy Abdelaziz, Assistant lecturer of family medicine, Sohag University
Other Study IDs: Soh-Med-25-2--3MD
Record Dates: First submitted 2025-02-12; First posted 2025-02-18 (Actual); Last update posted 2025-02-18 (Actual); Status verified 2025-02

CONDITIONS: Polycystic Ovary Syndrome (PCOS) Women
Keywords: PCOS; Quality of life; PCOSQ; BMI
MeSH Terms: conditions — Polycystic Ovary Syndrome

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Women with Polycystic ovary syndrome: women with PCOS visiting Gynecology and clinical nutrition outpatient clinics at Sohag university hospital
  Inclusion criteria:
  * Female cases between 18 and 45.
  * Females diagnosed with PCOS per Rotterdam criteria , the most commonly accepted and used for PCOS, a diagnosis is confirmed if any two of the three features (hyperandrogenism, oligomenorrhea or anovulation, and polycystic ovaries) are present in a woman of reproductive age[7].
  Exclusion criteria:
  * Females below 18 years old.
  * Females above 45 years old.
  * Patients having major life event or problem also affecting quality of life.

SUMMARY:
It is well-established that PCOS women suffer from anxiety, depression, and markedly reduced QoL ,but There has not yet been a nationally representative study to evaluate the PCOS health related Qol and factors affecting it among women in Egypt. So here we try to cover this gap in this study that will be designed to record the QOL of women with PCOS and factors affecting it.

This study aims to assess the health related quality of life of polycystic ovary syndrome and determine factors affecting the HRQOL

ELIGIBILITY:
Inclusion Criteria:

* • Female cases between 18 and 45.

  * Females diagnosed with PCOS per Rotterdam criteria , the most commonly accepted and used for PCOS, a diagnosis is confirmed if any two of the three features (hyperandrogenism, oligomenorrhea or anovulation, and polycystic ovaries) are present in a woman of reproductive age

Exclusion Criteria:

* • Females below 18 years old.

  * Females above 45 years old.
  * Patients having major life event or problem also affecting quality of life.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: women with PCOS visiting Gynecology and clinical nutrition outpatient clinics at Sohag university hospital during the period of 6 months.
Sampling Method: Probability Sample
Enrollment: 352 (Estimated)
Dates: Start 2025-03 (Estimated); Primary Completion 2025-09-01 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
health related quality of life of women with PCOS | 2 months after answering the polycystic ovary syndrome questionnaire
  The quality of life of the participants will be studied using Polycystic Ovary Syndrome Questionnaire (PCOSQ), which consists of 26 questions and 5 domains ,including emotions (eight questions), body hair (five questions), weight (five questions), infertility (four questions), and menstrual problems (four questions)

SECONDARY OUTCOMES:
Factors affecting health related quality of life of women with PCOS | 2 months after collecting data from the medical chart
  by medical chart developed by the investigator and the supervisors that will include Socio-demographic data of the women with PCOS, medical history and body measurements.

CONTACTS AND LOCATIONS:
Locations (1):
- faculty of medicine Sohag university, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Undecided